CLINICAL TRIAL: NCT01380093
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, 3-Way Crossover Study to Determine the Abuse Potential of Oral Administration of Crushed EMBEDA Relative to Crushed Controlled-Release Morphine Sulfate and Placebo in Non Dependent, Recreational Opioid Users
Brief Title: Abuse Potential of Orally Administered Crushed Embeda Compared to Crushed Controlled-Release Morphine and Placebo in Non-Dependent Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ALO-01-10-4005; B4541003
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2012-05-31 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2011-09

CONDITIONS: Nondependent Opioid Abuse, Episodic
Keywords: abuse potential; abuse liability; recreational opioid use; morphine
MeSH Terms: conditions — Recurrence | interventions — Morphine; morphine, naltrexone combination; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- MS Contin (morphine sulfate, controlled release) (Active Comparator)
  Interventions: Drug: MS Contin (morphine sulfate, controlled release)
- EMBEDA (morphine sulfate / naltrexone hydrochloride) (Experimental)
  Interventions: Drug: EMBEDA (morphine sulfate / naltrexone hydrochloride)

INTERVENTIONS:
Drug: Placebo — Single-dose, 2 x microcrystalline cellulose (weighed to equal weights of average tablet/capsule of active comparator) mixed with 150 ml artificially sweetened, non-carbonated beverage
  Arms: Placebo
Drug: MS Contin (morphine sulfate, controlled release) — Single-dose, 2 x 60 mg morphine sulfate whole tablets manually crushed and mixed with 150 ml artificially sweetened, non-carbonated beverage
  Arms: MS Contin (morphine sulfate, controlled release)
Drug: EMBEDA (morphine sulfate / naltrexone hydrochloride) — Single-dose, solution 2 x 60 mg morphine sulfate with sequestered 2.4 mg Naltrexone hydrochloride whole capsules manually crushed and mixed with 150 ml artificially sweetened, non-carbonated beverage
  Arms: EMBEDA (morphine sulfate / naltrexone hydrochloride)

SUMMARY:
The primary purpose of this study is to determine the abuse potential of EMBEDA compared to controlled release morphine when crushed and taken orally by non-dependent recreational opioid users; secondary purposes include to determine the abuse potential of crushed EMBEDA relative to placebo and and to compare the pharmacokinetics and safety of crushed EMBEDA with crushed controlled-release morphine and crushed placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a recreational opioid user who is NOT physically dependent on opioids based on Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition-Text Revision (DSM-IV-TR) criteria, and the Naloxone Challenge. A recreational opioid user is defined as recreationally abusing opioids for non-therapeutic purposes (i.e., for psychoactive effects) on at least 10 occasions within the last year and at least once in the 12 weeks prior to Visit 1.
* Subject is in generally good health as determined by medical history, physical examination, vital signs, clinical laboratory tests, and 12-lead electrocardiogram (ECG).

Exclusion Criteria:

* Has a history or current diagnosis of substance dependence (excluding caffeine and nicotine), as assessed by the Investigator using the DSM IV-TR criteria.
* Has participated in, is currently participating in, or is seeking treatment for substance- and/or alcohol-related disorders (excluding nicotine and caffeine).
* History or presence of any clinically significant illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, musculoskeletal, or psychiatric) or any other condition, which in the opinion of the Investigator would jeopardize the safety of the subject or the validity of the study results.
* Has a known allergy or history of hypersensitivity to morphine sulfate, opioids in general, naltrexone hydrochloride (HCl) or similar compounds and/or the known excipients in the investigational drug products.
* Has any condition in which an opioid is contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, or is suspected of having paralytic ileus).
* Females who are pregnant, lactating, or are planning to become pregnant during the course of the study. Females with a positive serum pregnancy test at Visit 1 or at any subsequent study visit will be excluded from participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Setnik B, Sommerville K, Goli V, Han L, Webster L. Assessment of pharmacodynamic effects following oral administration of crushed morphine sulfate and naltrexone hydrochloride extended-release capsules compared with crushed morphine sulfate controlled-release tablets and placebo in nondependent recreational opioid users. Pain Med. 2013 Aug;14(8):1173-86. doi: 10.1111/pme.12148. Epub 2013 Jun 7. PMID 23745947
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=ALO-01-10-4005&StudyName=Abuse%20Potential%20of%20Orally%20Administered%20Crushed%20Embeda%20Compared%20to%20Crushed%20Controlled-Release%20Morphine%20and%20Placebo%20in%20Non-Dependent%20Recre

RESULTS

PARTICIPANT FLOW:
Groups:
- Naloxone: Naloxone hydrochloride 0.2 milligram (mg) intravenously (IV) followed by additional 0.6 mg naloxone hydrochloride IV, each dose followed by an assessment for signs of withdrawal. Participants in this group were assigned to either morphine then placebo or placebo then morphine in the drug discrimination phase of the study.
- Morphine Then Placebo: Single dose of morphine sulfate 120 mg solution orally on Day 1 followed by single dose of matching placebo solution orally on Day 2. Participants in this group were assigned to morphine, placebo and EMBEDA in either of the 6 sequences in the treatment phase of the study.
- Placebo Then Morphine: Single dose of matching placebo solution orally on Day 1 followed by single dose of morphine sulfate 120 mg solution orally on Day 2. Participants in this group were assigned to morphine, placebo and EMBEDA in either of the 6 sequences in the treatment phase of the study.
- Placebo Then EMBEDA Then Morphine: Single dose of matching placebo solution orally in first intervention period; followed by single dose of solution of EMBEDA extended release (ER) capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in second intervention period; then single dose of solution of morphine sulfate (MS Contin) controlled release (CR) tablet 120 mg orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
- EMBEDA Then Morphine Then Placebo: Single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in first intervention period; followed by single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in second intervention period; then single dose of matching placebo solution orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
- Morphine Then Placebo Then EMBEDA: Single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in first intervention period; followed by single dose of matching placebo solution orally in second intervention period; then single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
- Morphine Then EMBEDA Then Placebo: Single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in first intervention period; followed by single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in second intervention period; then single dose of matching placebo solution orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
- Placebo Then Morphine Then EMBEDA: Single dose of matching placebo solution orally in first intervention period; followed by single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in second intervention period; then single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
- EMBEDA Then Placebo Then Morphine: Single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in first intervention period; followed by single dose of matching placebo solution orally in second intervention period; then single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in third intervention period. A washout period of at least 4 days (not exceeding 14 days) was maintained between each intervention period.
Period: Naloxone Challenge Phase
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 80 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TREATED | 59 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 59 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Screen failures | 21 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 1
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 30 | 29 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 29 | 29 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discrimination failure | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Drug Discrimination Phase: Day 2
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 29 | 29 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 20 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 9 | 13 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discrimination failure | 0 | 4 | 9 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Positive urine drug screen | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Backup participant | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: First Intervention
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Second Intervention
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 0 | 0 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 5 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Washout Period
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 0 | 0 | 5 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 5 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Phase: Third Intervention
Arm/Group | Naloxone | Morphine Then Placebo | Placebo Then Morphine | Placebo Then EMBEDA Then Morphine | EMBEDA Then Morphine Then Placebo | Morphine Then Placebo Then EMBEDA | Morphine Then EMBEDA Then Placebo | Placebo Then Morphine Then EMBEDA | EMBEDA Then Placebo Then Morphine
Started | 0 | 0 | 0 | 5 | 6 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 5 | 6 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non-compliance | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes all participants enrolled in the study.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 24.7 (4.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hours (hrs) (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: The evaluable population included all randomized participants who completed all 3 treatment periods of the treatment phase, contributed post-dose pharmacodynamic (PD) data from each period and did not have major protocol violations.
Measure: Mean (Standard Deviation); unit: hrs*mm
Groups:
- Placebo: Single dose of matching placebo solution orally in either of the first to third intervention periods.
- EMBEDA: Single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in either of the first to third intervention periods.
- Morphine: Single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in either of the first to third intervention periods.
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 88.3 (4.41) [83.6 to 93.6] | 100.3 (12.29) [95.5 to 105.5] | 124.7 (22.70) [120.4 to 130.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Least square (LS) mean and 95% confidence interval (CI) were calculated using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment. At least one primary outcome for each of drug liking and high was required to be significant with adjusted p-value less than or equal to 0.05; LS Mean Difference = -24.9, 95% CI 2-sided [-31.7 to -18.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; LS mean and 95% CI were calculated using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 11.9, 95% CI 2-sided [5.1 to 18.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 36.8, 95% CI 2-sided [30.0 to 43.6]

2. Primary Outcome: Drug Liking: Peak Effect (Emax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: The evaluable population included all randomized participants who completed all 3 treatment periods of the treatment phase, contributed post-dose PD data from each period and did not have major protocol violations.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 51.6 (4.21) [48.3 to 55.1] | 65.2 (11.21) [61.7 to 68.6] | 80.6 (13.09) [77.4 to 84.3]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; LS mean and 95% CI were calculated using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence. Planned power of at least 89% assumed a mean difference of 15 to 30 points and a standard deviation of paired differences of 15 to 20 points, with conservative multiple comparison adjustment for alpha of 0.025; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -15.7, 95% CI 2-sided [-20.2 to -11.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 13.4, 95% CI 2-sided [8.9 to 18.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 29.1, 95% CI 2-sided [24.6 to 33.7]

3. Primary Outcome: High: Area Under Effect Curve (AUE) From 0-2 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 2.0 (7.34) [-6.3 to 11.5] | 26.9 (27.72) [18.3 to 36.0] | 77.5 (34.40) [69.4 to 87.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -51.1, 95% CI 2-sided [-61.2 to -41.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 24.6, 95% CI 2-sided [14.5 to 34.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 75.7, 95% CI 2-sided [65.6 to 85.8]

4. Secondary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 37.8 (1.82) [35.7 to 40.2] | 43.1 (6.11) [40.9 to 45.4] | 51.8 (10.12) [49.8 to 54.3]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; LS mean, 95% CI, and unadjusted p-value were calculated using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -8.9, 95% CI 2-sided [-11.8 to -6.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 5.2, 95% CI 2-sided [2.3 to 8.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 14.1, 95% CI 2-sided [11.2 to 17.0]

5. Secondary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 188.6 (7.56) [179.1 to 199.1] | 217.9 (24.72) [208.1 to 228.2] | 265.6 (44.44) [256.9 to 276.9]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -48.8, 95% CI 2-sided [-62.0 to -35.5]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 29.0, 95% CI 2-sided [15.8 to 42.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 77.8, 95% CI 2-sided [64.5 to 91.0]

6. Secondary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 390.3 (15.19) [368.4 to 411.1] | 447.3 (60.82) [424.9 to 467.6] | 514.4 (87.10) [493.4 to 536.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -68.6, 95% CI 2-sided [-95.0 to -42.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 56.5, 95% CI 2-sided [30.1 to 82.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 125.1, 95% CI 2-sided [98.7 to 151.5]

7. Secondary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 591.0 (20.36) [560.2 to 619.4] | 658.2 (81.77) [626.7 to 685.9] | 732.9 (122.81) [702.7 to 761.9]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = -76.0, 95% CI 2-sided [-112.8 to -39.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = 66.5, 95% CI 2-sided [29.8 to 103.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 142.5, 95% CI 2-sided [105.7 to 179.3]

8. Secondary Outcome: Drug Liking: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1192.1 (29.73) [1150.1 to 1230.7] | 1263.0 (101.88) [1220.0 to 1300.5] | 1348.2 (174.53) [1306.1 to 1386.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS Mean Difference = -86.2, 95% CI 2-sided [-136.5 to -35.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0071, Mixed Models Analysis; LS Mean Difference = 69.8, 95% CI 2-sided [19.7 to 120.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 156.0, 95% CI 2-sided [105.7 to 206.3]

9. Secondary Outcome: Drug Liking: Time to Maximum (Peak) Effect (TEmax)
Description: Drug liking assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 5.8 (6.83) [3.8 to 7.5] | 4.8 (5.74) [2.8 to 6.5] | 2.7 (2.63) [0.7 to 4.5]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1254, Mixed Models Analysis; LS Mean Difference = 2.0, 95% CI 2-sided [-0.6 to 4.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4592, Mixed Models Analysis; LS Mean Difference = -1.0, 95% CI 2-sided [-3.6 to 1.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0251, Mixed Models Analysis; LS Mean Difference = -3.0, 95% CI 2-sided [-5.6 to -0.4]

10. Secondary Outcome: High: Area Under Effect Curve (AUE) From 0-1 Hour
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.9 (2.87) [-2.9 to 5.2] | 10.3 (12.26) [6.3 to 14.5] | 25.5 (16.26) [21.7 to 29.9]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -15.4, 95% CI 2-sided [-19.9 to -11.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 9.3, 95% CI 2-sided [4.8 to 13.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 24.7, 95% CI 2-sided [20.3 to 29.1]

11. Secondary Outcome: High: Area Under Effect Curve (AUE) From 0-4 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.4 (13.28) [-12.5 to 21.9] | 63.6 (53.04) [47.2 to 81.7] | 178.9 (64.56) [163.2 to 197.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -116.1, 95% CI 2-sided [-136.5 to -95.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 59.7, 95% CI 2-sided [39.3 to 80.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 175.8, 95% CI 2-sided [155.4 to 196.2]

12. Secondary Outcome: High: Area Under Effect Curve (AUE) From 0-8 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 6.5 (23.15) [-23.1 to 39.2] | 129.5 (101.43) [99.4 to 161.6] | 330.5 (109.02) [301.5 to 363.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -202.2, 95% CI 2-sided [-239.0 to -165.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 122.5, 95% CI 2-sided [85.7 to 159.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 324.6, 95% CI 2-sided [287.7 to 361.5]

13. Secondary Outcome: High: Area Under Effect Curve (AUE) From 0-12 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 8.1 (28.80) [0 to 49.8] | 160.7 (129.72) [121.5 to 201.7] | 412.3 (142.08) [374.4 to 454.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -253.0, 95% CI 2-sided [-301.5 to -204.5]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 151.9, 95% CI 2-sided [103.5 to 200.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 404.9, 95% CI 2-sided [356.4 to 453.3]

14. Secondary Outcome: High: Area Under Effect Curve (AUE) From 0-24 Hours
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 10.7 (35.41) [-39.6 to 65.1] | 180.3 (149.07) [129.0 to 233.8] | 485.4 (204.51) [435.7 to 540.6]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -306.8, 95% CI 2-sided [-370.9 to -242.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 168.6, 95% CI 2-sided [104.7 to 232.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 475.4, 95% CI 2-sided [411.3 to 539.6]

15. Secondary Outcome: High: Time to Maximum (Peak) Effect (TEmax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.8 (0.99) [0.1 to 1.3] | 2.7 (1.94) [2.1 to 3.3] | 2.5 (1.94) [1.9 to 3.1]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5607, Mixed Models Analysis; LS Mean Difference = 0.2, 95% CI 2-sided [-0.6 to 1.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 2.0, 95% CI 2-sided [1.2 to 2.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 1.8, 95% CI 2-sided [1.0 to 2.6]

16. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.8 (2.47) [-3.5 to 5.5] | 12.2 (13.74) [7.8 to 16.7] | 27.2 (17.64) [23.0 to 32.0]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -15.3, 95% CI 2-sided [-20.3 to -10.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 11.2, 95% CI 2-sided [6.3 to 16.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.5, 95% CI 2-sided [21.5 to 31.5]

17. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.8 (6.69) [-7.4 to 12.2] | 30.4 (29.84) [20.9 to 40.5] | 77.4 (38.39) [68.6 to 88.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -47.7, 95% CI 2-sided [-59.5 to -35.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 28.3, 95% CI 2-sided [16.5 to 40.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 76.0, 95% CI 2-sided [64.2 to 87.8]

18. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.1 (12.35) [-14.8 to 23.5] | 70.5 (58.34) [52.2 to 90.5] | 178.5 (73.28) [161.4 to 199.7]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -109.3, 95% CI 2-sided [-132.9 to -85.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 67.0, 95% CI 2-sided [43.5 to 90.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 176.3, 95% CI 2-sided [152.6 to 199.9]

19. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 6.2 (22.44) [-28.8 to 42.5] | 141.2 (120.31) [105.9 to 177.2] | 330.0 (122.85) [296.6 to 368.0]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -190.8, 95% CI 2-sided [-234.2 to -147.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 134.7, 95% CI 2-sided [91.5 to 178.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 325.5, 95% CI 2-sided [282.1 to 368.9]

20. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 7.8 (28.24) [0 to 53.9] | 174.6 (153.23) [129.0 to 220.4] | 417.4 (158.39) [373.8 to 465.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -244.9, 95% CI 2-sided [-302.0 to -187.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 166.5, 95% CI 2-sided [109.5 to 223.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 411.4, 95% CI 2-sided [354.3 to 468.6]

21. Secondary Outcome: Good Effects: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 10.2 (34.73) [-47.8 to 70.1] | 196.0 (176.48) [137.4 to 255.3] | 503.8 (223.88) [447.3 to 565.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -310.0, 95% CI 2-sided [-384.5 to -235.5]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 185.2, 95% CI 2-sided [110.8 to 259.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 495.1, 95% CI 2-sided [420.6 to 569.7]

22. Secondary Outcome: Good Effects: Peak Effect (Emax)
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 1.8 (5.38) [-4.6 to 8.6] | 32.6 (23.74) [26.2 to 39.4] | 63.0 (20.71) [56.7 to 69.9]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -30.5, 95% CI 2-sided [-38.7 to -22.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 30.8, 95% CI 2-sided [22.6 to 39.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 61.3, 95% CI 2-sided [53.1 to 69.5]

23. Secondary Outcome: Good Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Good effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.7 (0.99) [0.0 to 1.4] | 2.5 (2.13) [1.8 to 3.3] | 2.6 (2.47) [1.9 to 3.3]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.8671, Mixed Models Analysis; LS Mean Difference = -0.1, 95% CI 2-sided [-1.0 to 0.8]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = 1.8, 95% CI 2-sided [0.9 to 2.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 1.9, 95% CI 2-sided [1.0 to 2.8]

24. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.8 (2.23) [-2.8 to 4.9] | 9.8 (12.17) [6.0 to 13.7] | 22.6 (14.89) [19.0 to 26.7]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.0, 95% CI 2-sided [-17.0 to -9.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 8.8, 95% CI 2-sided [4.8 to 12.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 21.8, 95% CI 2-sided [17.8 to 25.8]

25. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.8 (6.41) [-6.2 to 11.3] | 26.7 (28.59) [18.4 to 35.9] | 71.5 (33.15) [63.7 to 81.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -45.3, 95% CI 2-sided [-55.3 to -35.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 24.5, 95% CI 2-sided [14.6 to 34.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 69.8, 95% CI 2-sided [59.9 to 79.8]

26. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.2 (11.95) [-12.2 to 21.8] | 63.8 (54.35) [47.9 to 81.9] | 172.2 (62.60) [156.9 to 191.0]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -109.1, 95% CI 2-sided [-129.3 to -88.8]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 60.1, 95% CI 2-sided [39.9 to 80.4]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 169.2, 95% CI 2-sided [148.9 to 189.5]

27. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 6.4 (22.45) [-21.4 to 38.4] | 125.6 (94.76) [97.3 to 157.1] | 331.8 (105.57) [304.3 to 364.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -207.0, 95% CI 2-sided [-242.0 to -172.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 118.7, 95% CI 2-sided [83.9 to 153.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 325.8, 95% CI 2-sided [290.8 to 360.7]

28. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 7.8 (27.85) [0 to 48.2] | 155.4 (117.10) [119.3 to 195.2] | 422.5 (136.00) [387.5 to 463.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -268.2, 95% CI 2-sided [-313.2 to -223.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 147.0, 95% CI 2-sided [102.1 to 191.9]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 415.2, 95% CI 2-sided [370.2 to 460.2]

29. Secondary Outcome: Any Effects: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 10.2 (33.80) [-36.0 to 62.7] | 176.4 (130.79) [129.6 to 228.3] | 510.8 (194.67) [465.6 to 564.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -336.0, 95% CI 2-sided [-395.4 to -276.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 165.6, 95% CI 2-sided [106.4 to 224.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 501.6, 95% CI 2-sided [442.2 to 561.0]

30. Secondary Outcome: Any Effects: Peak Effect (Emax)
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 1.9 (5.35) [-3.3 to 8.1] | 28.7 (20.03) [23.3 to 34.8] | 62.4 (18.59) [57.1 to 68.5]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -33.8, 95% CI 2-sided [-40.7 to -26.8]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.7, 95% CI 2-sided [19.7 to 33.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 60.4, 95% CI 2-sided [53.4 to 67.4]

31. Secondary Outcome: Any Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Any effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.8 (0.99) [0.1 to 1.4] | 3.1 (2.34) [2.5 to 3.8] | 2.8 (2.03) [2.0 to 3.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3345, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-0.4 to 1.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 2.4, 95% CI 2-sided [1.5 to 3.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 2.0, 95% CI 2-sided [1.1 to 2.8]

32. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.3 (0.92) [-0.4 to 1.1] | 0.6 (1.24) [-0.1 to 1.4] | 1.5 (3.70) [0.9 to 2.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0453, Mixed Models Analysis; LS Mean Difference = -1.0, 95% CI 2-sided [-2.0 to -0.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5637, Mixed Models Analysis; LS Mean Difference = 0.3, 95% CI 2-sided [-0.7 to 1.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0110, Mixed Models Analysis; LS Mean Difference = 1.3, 95% CI 2-sided [0.3 to 2.3]

33. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.5 (1.65) [-1.9 to 3.5] | 2.6 (4.40) [0.2 to 5.5] | 7.4 (12.50) [5.1 to 10.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0041, Mixed Models Analysis; LS Mean Difference = -4.9, 95% CI 2-sided [-8.2 to -1.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2178, Mixed Models Analysis; LS Mean Difference = 2.1, 95% CI 2-sided [-1.2 to 5.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 7.0, 95% CI 2-sided [3.7 to 10.3]

34. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.9 (3.20) [-6.0 to 9.3] | 7.7 (13.27) [0.9 to 16.2] | 27.1 (36.06) [20.3 to 35.6]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = -19.4, 95% CI 2-sided [-28.8 to -9.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1510, Mixed Models Analysis; LS Mean Difference = 6.9, 95% CI 2-sided [-2.6 to 16.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 26.2, 95% CI 2-sided [16.8 to 35.7]

35. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.6 (5.84) [-14.0 to 20.9] | 19.7 (37.56) [4.5 to 39.4] | 74.6 (80.92) [59.7 to 94.6]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -55.2, 95% CI 2-sided [-75.9 to -34.4]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0796, Mixed Models Analysis; LS Mean Difference = 18.5, 95% CI 2-sided [-2.2 to 39.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 73.6, 95% CI 2-sided [52.9 to 94.4]

36. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 2.1 (7.82) [0 to 30.2] | 28.4 (56.67) [6.4 to 57.1] | 110.3 (116.60) [89.2 to 140.0]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -82.8, 95% CI 2-sided [-112.9 to -52.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0780, Mixed Models Analysis; LS Mean Difference = 26.9, 95% CI 2-sided [-3.1 to 56.9]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 109.7, 95% CI 2-sided [79.6 to 139.8]

37. Secondary Outcome: Bad Effects: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.6 (13.62) [-27.7 to 41.7] | 36.8 (76.50) [6.2 to 75.6] | 147.2 (157.74) [118.1 to 187.6]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -111.9, 95% CI 2-sided [-153.7 to -70.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1089, Mixed Models Analysis; LS Mean Difference = 33.9, 95% CI 2-sided [-7.8 to 75.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 145.8, 95% CI 2-sided [104.1 to 187.5]

38. Secondary Outcome: Bad Effects: Peak Effect (Emax)
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 0.6 (1.60) [-3.4 to 5.4] | 6.6 (10.30) [2.6 to 11.4] | 20.1 (18.98) [16.3 to 25.1]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.7, 95% CI 2-sided [-18.8 to -8.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0215, Mixed Models Analysis; LS Mean Difference = 6.0, 95% CI 2-sided [0.9 to 11.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.7, 95% CI 2-sided [14.6 to 24.8]

39. Secondary Outcome: Bad Effects: Time to Maximum (Peak) Effect (TEmax)
Description: Bad effects VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.9 (1.60) [0.1 to 1.9] | 2.2 (2.38) [1.4 to 3.2] | 4.5 (3.56) [3.7 to 5.5]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; LS Mean Difference = -2.3, 95% CI 2-sided [-3.6 to -1.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0455, Mixed Models Analysis; LS Mean Difference = 1.3, 95% CI 2-sided [0.0 to 2.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 3.6, 95% CI 2-sided [2.3 to 4.9]

40. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: Pre-dose, 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.4 (1.28) [0.0 to 1.0] | 0.5 (1.16) [0.0 to 1.1] | 0.8 (2.25) [0.3 to 1.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3749, Mixed Models Analysis; LS Mean Difference = -0.3, 95% CI 2-sided [-0.9 to 0.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7939, Mixed Models Analysis; LS Mean Difference = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2524, Mixed Models Analysis; LS Mean Difference = 0.4, 95% CI 2-sided [-0.3 to 1.0]

41. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: Pre-dose, 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.7 (1.73) [-0.9 to 2.7] | 2.1 (4.12) [0.4 to 4.1] | 3.7 (8.14) [2.1 to 5.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1211, Mixed Models Analysis; LS Mean Difference = -1.7, 95% CI 2-sided [-3.8 to 0.5]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1997, Mixed Models Analysis; LS Mean Difference = 1.4, 95% CI 2-sided [-0.7 to 3.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis; LS Mean Difference = 3.1, 95% CI 2-sided [0.9 to 5.2]

42. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.0 (2.78) [-4.1 to 7.4] | 5.5 (11.30) [0.5 to 11.9] | 15.3 (26.61) [10.3 to 21.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis; LS Mean Difference = -9.8, 95% CI 2-sided [-16.7 to -3.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1918, Mixed Models Analysis; LS Mean Difference = 4.5, 95% CI 2-sided [-2.3 to 11.4]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 14.4, 95% CI 2-sided [7.5 to 21.2]

43. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.6 (5.17) [-12.2 to 20.4] | 16.5 (39.86) [2.8 to 35.3] | 47.1 (75.02) [34.3 to 66.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis; LS Mean Difference = -31.5, 95% CI 2-sided [-50.2 to -12.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1136, Mixed Models Analysis; LS Mean Difference = 14.9, 95% CI 2-sided [-3.7 to 33.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 46.5, 95% CI 2-sided [27.8 to 65.1]

44. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 2.2 (7.42) [0.0 to 31.5] | 25.2 (61.13) [3.7 to 54.8] | 76.9 (119.64) [57.3 to 108.4]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; LS Mean Difference = -53.6, 95% CI 2-sided [-83.2 to -24.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1207, Mixed Models Analysis; LS Mean Difference = 23.2, 95% CI 2-sided [-6.3 to 52.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 76.8, 95% CI 2-sided [47.3 to 106.4]

45. Secondary Outcome: Nausea: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.8 (13.69) [-26.9 to 44.4] | 35.3 (76.53) [5.0 to 76.3] | 108.3 (171.22) [80.7 to 152.1]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = -75.8, 95% CI 2-sided [-118.6 to -33.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1410, Mixed Models Analysis; LS Mean Difference = 31.8, 95% CI 2-sided [-10.8 to 74.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 107.7, 95% CI 2-sided [64.9 to 150.5]

46. Secondary Outcome: Nausea: Peak Effect (Emax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 0.8 (2.41) [-2.5 to 5.3] | 5.2 (10.41) [1.8 to 9.6] | 14.9 (17.14) [11.8 to 19.6]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.0, 95% CI 2-sided [-14.4 to -5.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0529, Mixed Models Analysis; LS Mean Difference = 4.3, 95% CI 2-sided [-0.1 to 8.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 14.3, 95% CI 2-sided [9.9 to 18.7]

47. Secondary Outcome: Nausea: Time to Maximum (Peak) Effect (TEmax)
Description: Nausea VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 1.4 (4.17) [0.0 to 2.9] | 2.5 (4.69) [1.1 to 4.0] | 4.3 (3.52) [2.9 to 5.8]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0806, Mixed Models Analysis; LS Mean Difference = -1.8, 95% CI 2-sided [-3.8 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2769, Mixed Models Analysis; LS Mean Difference = 1.1, 95% CI 2-sided [-0.9 to 3.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0056, Mixed Models Analysis; LS Mean Difference = 2.9, 95% CI 2-sided [0.9 to 5.0]

48. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.3 (1.09) [-0.3 to 1.2] | 0.3 (0.86) [-0.3 to 1.1] | 1.0 (3.50) [0.4 to 1.9]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1100, Mixed Models Analysis; LS Mean Difference = -0.8, 95% CI 2-sided [-1.7 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.9421, Mixed Models Analysis; LS Mean Difference = 0, 95% CI 2-sided [-1.0 to 0.9]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1266, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [-0.2 to 1.7]

49. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.6 (1.75) [-1.3 to 3.1] | 1.7 (4.25) [-0.3 to 4.1] | 4.2 (10.19) [2.3 to 6.7]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0723, Mixed Models Analysis; LS Mean Difference = -2.6, 95% CI 2-sided [-5.3 to 0.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4515, Mixed Models Analysis; LS Mean Difference = 1.1, 95% CI 2-sided [-1.7 to 3.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0121, Mixed Models Analysis; LS Mean Difference = 3.6, 95% CI 2-sided [0.8 to 6.4]

50. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.0 (3.22) [-4.5 to 8.0] | 5.2 (12.28) [-0.3 to 12.2] | 16.1 (28.88) [10.6 to 23.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0059, Mixed Models Analysis; LS Mean Difference = -11.0, 95% CI 2-sided [-18.7 to -3.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2800, Mixed Models Analysis; LS Mean Difference = 4.2, 95% CI 2-sided [-3.5 to 11.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 15.1, 95% CI 2-sided [7.5 to 22.8]

51. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.7 (6.27) | 14.8 (35.83) | 50.7 (72.35)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = -36.7, 95% CI 2-sided [-54.8 to -18.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1488, Mixed Models Analysis; LS Mean Difference = 13.2, 95% CI 2-sided [-4.8 to 31.2]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 49.9, 95% CI 2-sided [31.8 to 67.9]

52. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 2.3 (8.53) | 22.5 (54.79) | 80.9 (113.22)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -60.1, 95% CI 2-sided [-88.5 to -31.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1556, Mixed Models Analysis; LS Mean Difference = 20.4, 95% CI 2-sided [-8.0 to 48.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 80.4, 95% CI 2-sided [52.0 to 108.9]

53. Secondary Outcome: Feel Sick: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.9 (14.72) | 31.1 (73.35) | 112.8 (160.44)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; LS Mean Difference = -84.0, 95% CI 2-sided [-124.8 to -43.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1826, Mixed Models Analysis; LS Mean Difference = 27.4, 95% CI 2-sided [-13.3 to 68.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 111.4, 95% CI 2-sided [70.6 to 152.2]

54. Secondary Outcome: Feel Sick: Peak Effect (Emax)
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 0.7 (1.96) | 4.9 (11.06) | 16.4 (17.38)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -11.7, 95% CI 2-sided [-16.4 to -7.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0811, Mixed Models Analysis; LS Mean Difference = 4.2, 95% CI 2-sided [-0.5 to 8.9]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 15.9, 95% CI 2-sided [11.1 to 20.6]

55. Secondary Outcome: Feel Sick: Time to Maximum (Peak) Effect (TEmax)
Description: Feel sick VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.9 (2.00) | 1.8 (2.77) | 4.3 (3.45)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; LS Mean Difference = -2.5, 95% CI 2-sided [-3.8 to -1.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1631, Mixed Models Analysis; LS Mean Difference = 1.0, 95% CI 2-sided [-0.4 to 2.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 3.4, 95% CI 2-sided [2.1 to 4.8]

56. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr(0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.4 (1.30) | 2.4 (6.57) | 3.6 (5.13)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2117, Mixed Models Analysis; LS Mean Difference = -1.2, 95% CI 2-sided [-3.1 to 0.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0345, Mixed Models Analysis; LS Mean Difference = 2.1, 95% CI 2-sided [0.2 to 4.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; LS Mean Difference = 3.3, 95% CI 2-sided [1.4 to 5.2]

57. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.7 (1.91) | 9.1 (12.63) | 21.3 (21.28)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = -12.2, 95% CI 2-sided [-18.4 to -6.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis; LS Mean Difference = 8.4, 95% CI 2-sided [2.3 to 14.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 20.6, 95% CI 2-sided [14.4 to 26.8]

58. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.7 (4.31) | 35.9 (38.78) | 74.2 (61.41)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -38.2, 95% CI 2-sided [-55.6 to -20.8]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 34.4, 95% CI 2-sided [17.0 to 51.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 72.6, 95% CI 2-sided [55.2 to 90.0]

59. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Groups:
- EMBEDA: Single dose of EMBEDA solution containing 120 mg morphine sulfate / 4.8 mg naltrexone hydrochloride administered orally in either of the first to third intervention periods.
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 4.2 (10.15) | 97.6 (103.13) | 199.2 (141.96)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -100.3, 95% CI 2-sided [-142.2 to -58.4]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 93.9, 95% CI 2-sided [52.1 to 135.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 194.2, 95% CI 2-sided [152.3 to 236.1]

60. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 5.3 (13.05) | 138.5 (140.93) | 287.5 (196.29)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -147.4, 95% CI 2-sided [-205.1 to -89.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 134.1, 95% CI 2-sided [76.5 to 191.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 281.5, 95% CI 2-sided [223.7 to 339.2]

61. Secondary Outcome: Sleepy: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 7.6 (21.06) | 175.5 (175.65) | 378.7 (267.76)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -201.4, 95% CI 2-sided [-279.3 to -123.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 169.1, 95% CI 2-sided [91.5 to 246.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 370.5, 95% CI 2-sided [292.7 to 448.4]

62. Secondary Outcome: Sleepy: Peak Effect (Emax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 1.5 (3.71) | 27.1 (22.75) | 43.9 (21.93)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -16.4, 95% CI 2-sided [-23.8 to -9.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.7, 95% CI 2-sided [18.3 to 33.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 42.1, 95% CI 2-sided [34.7 to 49.5]

63. Secondary Outcome: Sleepy: Time to Maximum (Peak) Effect (TEmax)
Description: Sleepy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 1.1 (2.20) | 4.0 (2.94) | 5.3 (2.81)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0253, Mixed Models Analysis; LS Mean Difference = -1.4, 95% CI 2-sided [-2.6 to -0.2]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 2.8, 95% CI 2-sided [1.6 to 4.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 4.2, 95% CI 2-sided [3.0 to 5.4]

64. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.4 (1.28) | 0.9 (2.41) | 3.0 (5.73)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0062, Mixed Models Analysis; LS Mean Difference = -2.1, 95% CI 2-sided [-3.7 to -0.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4998, Mixed Models Analysis; LS Mean Difference = 0.5, 95% CI 2-sided [-1.0 to 2.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; LS Mean Difference = 2.7, 95% CI 2-sided [1.1 to 4.2]

65. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.6 (1.70) | 2.8 (6.26) | 9.9 (15.14)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; LS Mean Difference = -7.0, 95% CI 2-sided [-11.1 to -3.0]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2693, Mixed Models Analysis; LS Mean Difference = 2.2, 95% CI 2-sided [-1.8 to 6.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 9.3, 95% CI 2-sided [5.3 to 13.3]

66. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.0 (2.93) | 9.5 (21.81) | 26.1 (41.05)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0042, Mixed Models Analysis; LS Mean Difference = -16.2, 95% CI 2-sided [-27.2 to -5.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1139, Mixed Models Analysis; LS Mean Difference = 8.7, 95% CI 2-sided [-2.2 to 19.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 25.0, 95% CI 2-sided [14.1 to 35.9]

67. Primary Outcome: High: Peak Effect (Emax)
Description: High VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 1.8 (5.73) [-3.7 to 8.1] | 29.2 (20.72) [23.6 to 35.3] | 64.1 (18.85) [58.5 to 70.2]
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -34.9, 95% CI 2-sided [-42.1 to -27.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 27.2, 95% CI 2-sided [20.1 to 34.4]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — p-value adjusted for multiple comparisons with Hochberg adjustment; LS Mean Difference = 62.1, 95% CI 2-sided [54.9 to 69.4]

68. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 1.7 (5.93) | 20.9 (51.17) | 56.7 (87.00)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0039, Mixed Models Analysis; LS Mean Difference = -35.1, 95% CI 2-sided [-58.5 to -11.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1026, Mixed Models Analysis; LS Mean Difference = 19.3, 95% CI 2-sided [-4.0 to 42.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 54.4, 95% CI 2-sided [31.0 to 77.8]

69. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 2.4 (8.68) | 27.4 (66.65) | 71.4 (111.82)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0051, Mixed Models Analysis; LS Mean Difference = -43.3, 95% CI 2-sided [-73.1 to -13.5]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0941, Mixed Models Analysis; LS Mean Difference = 25.3, 95% CI 2-sided [-4.4 to 55.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 68.6, 95% CI 2-sided [38.8 to 98.4]

70. Secondary Outcome: Dizzy: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 4.0 (14.73) | 36.0 (82.99) | 85.5 (135.09)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0083, Mixed Models Analysis; LS Mean Difference = -49.0, 95% CI 2-sided [-85.0 to -13.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0766, Mixed Models Analysis; LS Mean Difference = 32.3, 95% CI 2-sided [-3.5 to 68.1]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 81.3, 95% CI 2-sided [45.4 to 117.3]

71. Secondary Outcome: Dizzy: Peak Effect (Emax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). Emax = Maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 0.7 (2.45) | 5.5 (11.18) | 13.7 (17.66)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0018, Mixed Models Analysis; LS Mean Difference = -8.0, 95% CI 2-sided [-12.9 to -3.1]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0527, Mixed Models Analysis; LS Mean Difference = 4.8, 95% CI 2-sided [-0.1 to 9.7]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 12.8, 95% CI 2-sided [7.9 to 17.7]

72. Secondary Outcome: Dizzy: Time to Maximum (Peak) Effect (TEmax)
Description: Dizzy VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm). TEmax = Time to maximum observed score.
Time Frame: 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 0.5 (0.09) | 2.0 (2.57) | 2.4 (2.60)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.3986, Mixed Models Analysis; LS Mean Difference = -0.4, 95% CI 2-sided [-1.4 to 0.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0023, Mixed Models Analysis; LS Mean Difference = 1.5, 95% CI 2-sided [0.6 to 2.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; LS Mean Difference = 1.9, 95% CI 2-sided [1.0 to 2.9]

73. Secondary Outcome: Overall Drug Liking Effect at 24 Hours
Description: Overall drug liking VAS assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100 mm VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm= "neither like nor dislike", and 100 mm= "strong liking").
Time Frame: 24 hrs post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 50.6 (3.06) | 58.8 (17.68) | 69.8 (20.23)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis; LS Mean Difference = -11.2, 95% CI 2-sided [-18 to -4]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0286, Mixed Models Analysis; LS Mean Difference = 8.1, 95% CI 2-sided [1 to 15]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 19.3, 95% CI 2-sided [12 to 27]

74. Secondary Outcome: Take Drug Again Effect at 24 Hours
Description: Take drug again VAS is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely would not", 50 mm = "do not care", and 100 mm = "definitely would").
Time Frame: 24 hrs post dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 49.8 (4.41) | 58.0 (21.90) | 70.6 (24.53)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis; LS Mean Difference = -13.0, 95% CI 2-sided [-22 to -4]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0700, Mixed Models Analysis; LS Mean Difference = 8.2, 95% CI 2-sided [-1 to 17]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 21.2, 95% CI 2-sided [12 to 30]

75. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-1 Hour
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-1) = Area under the effect versus time curve from time 0 to 1 hr (0-1).
Time Frame: Pre-dose, 0.5 and 1 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.0 (0.40) | -0.5 (0.38) | -1.2 (0.60)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 0.7, 95% CI 2-sided [0.5 to 0.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -1.0]

76. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-2 Hours
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-2) = Area under the effect versus time curve from time 0 to 2 hrs (0-2).
Time Frame: Pre-dose, 0.5, 1, 1.5 and 2 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.0 (0.87) | -1.7 (1.07) | -4.1 (1.31)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 2.4, 95% CI 2-sided [1.9 to 2.9]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.7, 95% CI 2-sided [-2.2 to -1.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -4.1, 95% CI 2-sided [-4.6 to -3.6]

77. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-4 Hours
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-4) = Area under the effect versus time curve from time 0 to 4 hrs (0-4).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | -0.1 (1.67) | -5.4 (2.29) | -10.3 (2.58)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 4.9, 95% CI 2-sided [3.9 to 5.8]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -5.3, 95% CI 2-sided [-6.3 to -4.3]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -10.1, 95% CI 2-sided [-11.1 to -9.2]

78. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-8 Hours
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-8) = Area under the effect versus time curve from time 0 to 8 hrs (0-8).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.0 (3.25) | -13.8 (4.36) | -22.5 (5.35)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 8.6, 95% CI 2-sided [6.6 to 10.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -13.8, 95% CI 2-sided [-15.9 to -11.8]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -22.4, 95% CI 2-sided [-24.5 to -20.4]

79. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-12 Hours
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-12) = Area under the effect versus time curve from time 0 to 12 hrs (0-12).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 0.7 (4.78) | -20.8 (6.80) | -32.6 (7.95)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 11.7, 95% CI 2-sided [8.7 to 14.7]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -21.5, 95% CI 2-sided [-24.5 to -18.6]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -33.2, 95% CI 2-sided [-36.2 to -30.2]

80. Secondary Outcome: Pupillometry: Area Under Effect Curve (AUE) From 0-24 Hours
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. AUE (0-24) = Area under the effect versus time curve from time 0 to 24 hrs (0-24).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs*mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs*mm | 3.5 (9.19) | -34.2 (13.96) | -51.8 (15.26)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 17.5, 95% CI 2-sided [11.6 to 23.3]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -37.7, 95% CI 2-sided [-43.6 to -31.9]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -55.2, 95% CI 2-sided [-61.1 to -49.3]

81. Secondary Outcome: Pupillometry: Peak Effect (Emax)
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. Emax = Smallest post-dose pupil size.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
mm | 5.6 (0.76) | 3.9 (0.71) | 2.8 (0.74)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = 1.1, 95% CI 2-sided [0.8 to 1.4]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -1.8, 95% CI 2-sided [-2.1 to -1.5]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; LS Mean Difference = -2.9, 95% CI 2-sided [-3.2 to -2.6]

82. Secondary Outcome: Pupillometry: Time to Maximum (Peak) Effect (TEmax)
Description: Pupillometry assessments measured change in pupil size (miosis) as an indicator of opioid pharmacological properties. The same eye for each participant was used for all measurements during the study. Participants had the size of their pupil measured (in mm) using a pupillometer. Measurements were made in a dimly lit (mesopic) room with controlled lighting conditions. TEmax = Time to smallest post-dose pupil size.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Placebo | EMBEDA | Morphine
Number analyzed (Participants) | 33 | 33 | 33
hrs | 4.8 (6.83) | 5.6 (2.26) | 3.2 (1.64)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0262, Mixed Models Analysis; LS Mean Difference = 2.5, 95% CI 2-sided [0.3 to 4.6]
Statistical Analysis 2: Comparison: Placebo vs EMBEDA; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4180, Mixed Models Analysis; LS Mean Difference = 0.9, 95% CI 2-sided [-1.3 to 3.0]
Statistical Analysis 3: Comparison: Placebo vs Morphine; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.1479, Mixed Models Analysis; LS Mean Difference = -1.6, 95% CI 2-sided [-3.7 to 0.6]

83. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Morphine
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs | 0.9 (0.48) | 0.7 (0.25)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Tmax was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0181, Mixed Models Analysis; LS Mean Difference = 0.21, 90% CI 2-sided [0.07 to 0.35]

84. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Morphine
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
picogram/milliliter (pg/mL) | 79308.6 (31555.86) | 103621 (34005.3)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed Cmax was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Geometric mean ratio = 0.75, 90% CI 2-sided [0.68 to 0.83]

85. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-1)] of Morphine
Description: AUC (0-1) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-1).
Time Frame: Pre-dose, 0.5 and 1 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 52644.9 (19951.60) | 67920.1 (24702.80)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-1) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Geometric mean ratio = 0.77, 90% CI 2-sided [0.69 to 0.86]

86. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-2)] of Morphine
Description: AUC (0-2) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-2).
Time Frame: Pre-dose, 0.5, 1, 1.5 and 2 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 112989 (33784.6) | 129721 (39670.7)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-2) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; Geometric mean ratio = 0.86, 90% CI 2-sided [0.79 to 0.94]

87. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-4)] of Morphine
Description: AUC (0-4) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-4).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 197745 (54807.4) | 199442 (60559.8)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-4) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.6399, Mixed Models Analysis; Geometric mean ratio = 0.98, 90% CI 2-sided [0.91 to 1.06]

88. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-8)] of Morphine
Description: AUC (0-8) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-8).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 269743 (77664.5) | 263270 (76706.0)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-8) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.9057, Mixed Models Analysis; Geometric mean ratio = 1.00, 90% CI 2-sided [0.94 to 1.08]

89. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-12)] of Morphine
Description: AUC (0-12) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-12).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 303428 (86669.9) | 288324 (81697.4)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-12) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.4250, Mixed Models Analysis; Geometric mean ratio = 1.03, 90% CI 2-sided [0.97 to 1.10]

90. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] of Morphine
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero to time of last quantifiable concentration (0-24).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 376260 (104635.5) | 335357 (91242.6)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-24) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0204, Mixed Models Analysis; Geometric mean ratio = 1.10, 90% CI 2-sided [1.03 to 1.18]

91. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Morphine
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA | Morphine
Number analyzed (Participants) | 35 | 33
hrs*pg/mL | 551755 (476987.0) | 369270 (98821.5)
Statistical Analysis 1: Comparison: EMBEDA vs Morphine; Natural log transformed AUC (0-∞) was analyzed using linear mixed model with fixed effects for sequence, period and treatment, and a random effect for participant nested in sequence; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Geometric mean ratio = 1.32, 90% CI 2-sided [1.17 to 1.49]

92. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Naltrexone
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs | 0.8 (0.32)

93. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Naltrexone
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
pg/mL | 978.83 (713.748)

94. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-1)] of Naltrexone
Description: as for outcome 85
Time Frame: Pre-dose, 0.5 and 1 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 619.24 (441.602)

95. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-2)] of Naltrexone
Description: as for outcome 86
Time Frame: Pre-dose, 0.5, 1, 1.5 and 2 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 1270.91 (700.063)

96. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-4)] of Naltrexone
Description: as for outcome 87
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 2018.23 (1000.217)

97. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-8)] of Naltrexone
Description: as for outcome 88
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 2577.19 (1228.398)

98. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-12)] of Naltrexone
Description: as for outcome 89
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 2813.34 (1337.306)

99. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] of Naltrexone
Description: as for outcome 90
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 3159.91 (1522.915)

100. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Naltrexone
Description: as for outcome 91
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 3320.90 (1616.514)

101. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Naltrexone Metabolite (6-beta-naltrexol)
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs | 1.0 (0.61)

102. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Naltrexone Metabolite (6-beta-naltrexol)
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
pg/mL | 6226.3 (2158.29)

103. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-1)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 85
Time Frame: Pre-dose, 0.5 and 1 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 3934.5 (1529.66)

104. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-2)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 86
Time Frame: Pre-dose, 0.5, 1, 1.5 and 2 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 8916.1 (2747.62)

105. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-4)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 87
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3 and 4 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 16532.5 (4351.58)

106. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-8)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 88
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6 and 8 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 26634.5 (6167.97)

107. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-12)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 89
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 12 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 33324.9 (7309.76)

108. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-24)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 90
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 47809.1 (10184.33)

109. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Naltrexone Metabolite (6-beta-naltrexol)
Description: as for outcome 91
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hrs post-dose
Population: Safety population included all participants who received at least one dose of study drug in the Treatment Phase.
Measure: Mean (Standard Deviation); unit: hrs*pg/mL
Arm/Group | EMBEDA
Number analyzed (Participants) | 35
hrs*pg/mL | 74931.5 (25580.10)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Naloxone (Naloxone Challenge Phase): Naloxone hydrochloride 0.2 mg IV followed by additional 0.6 mg naloxone hydrochloride IV, each dose followed by an assessment for signs of withdrawal.
- Placebo (Drug Discrimination Phase): Single dose of matching placebo solution orally on Day 1 or 2.
- Morphine (Drug Discrimination Phase): Single dose of morphine sulfate 120 mg solution orally on Day 1 or 2.
- Placebo (Treatment Phase): Single dose of matching placebo solution orally in either of the first to third intervention periods.
- EMBEDA (Treatment Phase): Single dose of solution of EMBEDA ER capsule containing 120 mg morphine sulfate and 4.8 mg naltrexone hydrochloride orally in either of the first to third intervention periods.
- Morphine (Treatment Phase): Single dose of solution of morphine sulfate (MS Contin) CR tablet 120 mg orally in either of the first to third intervention periods.
Arm/Group | Naloxone (Naloxone Challenge Phase) | Placebo (Drug Discrimination Phase) | Morphine (Drug Discrimination Phase) | Placebo (Treatment Phase) | EMBEDA (Treatment Phase) | Morphine (Treatment Phase)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58 | 0/59 | 0/36 | 1/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/59 | 1/58 | 51/59 | 2/36 | 10/35 | 27/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxone (Naloxone Challenge Phase) (N=59) | Placebo (Drug Discrimination Phase) (N=58) | Morphine (Drug Discrimination Phase) (N=59) | Placebo (Treatment Phase) (N=36) | EMBEDA (Treatment Phase) (N=35) | Morphine (Treatment Phase) (N=33)
Bipolar Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Schizoaffective Disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Naloxone (Naloxone Challenge Phase) (N=59) | Placebo (Drug Discrimination Phase) (N=58) | Morphine (Drug Discrimination Phase) (N=59) | Placebo (Treatment Phase) (N=36) | EMBEDA (Treatment Phase) (N=35) | Morphine (Treatment Phase) (N=33)
Nausea (Gastrointestinal disorders) | 0 | 0 | 36 | 1 | 3 | 15
Vomiting (Gastrointestinal disorders) | 0 | 0 | 27 | 0 | 0 | 14
Dizziness (Nervous system disorders) | 0 | 0 | 11 | 0 | 2 | 6
Somnolence (Nervous system disorders) | 0 | 0 | 10 | 0 | 4 | 3
Headache (Nervous system disorders) | 0 | 1 | 4 | 1 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 24 | 0 | 2 | 12
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0 | 2 | 3
Pain (General disorders) | 0 | 0 | 3 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.